CLINICAL TRIAL: NCT06106880
Title: Alleviation of Upper Respiratory Inflammation and Associated Common Cold Symptoms
Brief Title: Alleviation of Common Cold Symptoms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Biological Laboratories Inc (Other)
Collaborators: Econometrica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro 00048530
Record Dates: First submitted 2023-10-18; First posted 2023-10-30 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Common Cold; Pharyngitis; Fever; Congestion; Rhinorrhea; Cough; Sore-throat; Sore Throats Viral; Malaise; Headache; Runny Nose; Sneezing
Keywords: Common Cold; Pharyngitis; Fever; Congestion; Rhinorrhea; Cough; Sore Throat; Malaise; Headache; Runny Nose; Sneezing; Inflammation
MeSH Terms: conditions — Common Cold; Pharyngitis; Fever; Rhinorrhea; Cough; Headache; Sneezing; Inflammation | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A: Placebo Throat Spray and Placebo Tablet (Placebo Comparator): The placebo spray contained vehicle buffer, a sub-therapeutic dose of menthol, and a sweetener.
  Placebo Tablet: Looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Interventions: Other: Placebo Throat Spray and Placebo Tablet
- Group B: Wintergreen Throat Spray and Aspirin Tablet (Active Comparator): The liquid spray contained wintergreen oil, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  Aspirin in a 325mg tablet
  Interventions: Drug: Wintergreen Throat Spray and Aspirin Tablet
- Group C: Aspirin Throat Spray and Placebo Tablet (Active Comparator): The liquid spray contained 6mg dissolved acetyl salicylic acid per dose, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  Placebo Tablet: Looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Interventions: Drug: Aspirin Throat Spray and Placebo Tablet
- Group D: Wintergreen Throat Spray and Placebo Tablet (Active Comparator): The liquid spray contained wintergreen oil, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  Placebo Tablet: Looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Interventions: Dietary Supplement: Wintergreen Throat Spray and Placebo Tablet

INTERVENTIONS:
Drug: Wintergreen Throat Spray and Aspirin Tablet — The liquid spray contained wintergreen oil, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  Aspirin in a 325mg tablet
  Other Names: Group B
  Arms: Group B: Wintergreen Throat Spray and Aspirin Tablet
Drug: Aspirin Throat Spray and Placebo Tablet — The liquid spray contained 6mg dissolved acetyl salicylic acid per dose, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  Placebo Tablet: Looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Other Names: Group C
  Arms: Group C: Aspirin Throat Spray and Placebo Tablet
Dietary Supplement: Wintergreen Throat Spray and Placebo Tablet — The liquid spray contained wintergreen oil, menthol, lactoferrin, lysozyme, aloe, and glycerin.
  The placebo tablet looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Other Names: Group D
  Arms: Group D: Wintergreen Throat Spray and Placebo Tablet
Other: Placebo Throat Spray and Placebo Tablet — The placebo spray contained vehicle buffer, a sub-therapeutic dose of menthol, and a sweetener.
  The placebo tablet looked like the treatment aspirin tablet but contained no drug and only inactive excipients.
  Other Names: Group A
  Arms: Group A: Placebo Throat Spray and Placebo Tablet

SUMMARY:
Upper respiratory infections (URIs) have long posed a significant burden to the US healthcare system. Well before the coronavirus disease of 2019 (COVID-19) pandemic they have been among the most common acute outpatient illnesses, causing 75-100 million physician visits each year on average, and costing the health care system billions of dollars annually. This double-blind randomized placebo-controlled study tested the efficacy of two anti-inflammatory throat sprays against placebo and against a throat spray taken in conjunction with 325mg of aspirin, a well-known systemically administered cyclooxygenase (COX) inhibitor. Participants having common cold symptoms lasting less than two days were enrolled and given treatment to administer at home. Various common cold symptoms were assessed and measured via clinically validated self-assessment scales. Participants were screened for influenza and COVID-19 before enrollment and were excluded if found positive.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy adults with cold symptoms including sore throat who do not meet any of the exclusion criteria listed below,
* who rate their sore throat at least a 3 on a 10-point scale,
* who have had a sore throat for less than 48 hours by the time they complete the intake clinical trial manager (CTM) assessment.

Exclusion Criteria:

* Sore throat for more than 2 full days at the time of intake CTM assessment
* Fever or development of fever during the course of the trial
* Positive COVID-19 test or influenza test at clinical trial administrator (CTA) visit
* Likelihood of strep throat (to be determined by physician PI to the best of their ability)
* Less than 2 doses of the coronavirus (COVID-19) vaccine
* Any allergies to eggs, milk, or aspirin
* Females who are pregnant or test positive for pregnancy at the CTA visit
* Any chronic disease such as asthma, hypertension, post-nasal drip, gastroesophageal reflux disease (GERD), cardiopulmonary obstructive disorder (COPD), diabetes, cancer, HIV
* Any history of allergy in the last 14 days for which they took medication
* Anyone with fever above 101 or who has taken medication other than birth control in the last 30 days
* Anyone taking an Angiotensin Converting Enzyme (ACE) inhibitor
* Participation in another clinical trial within the last 6 months or during this trial
* Anyone who smokes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2023-04-08 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Relief of Sore Throat Pain | 36 hours
  A time-weighted summed difference in pain intensity on the sore throat pain intensity scale (STPIS) after the first dose of medication (STPIS 1st entry Day 1 compared to STPIS 4th entry Day 2). On the STPIS, 0mm, the leftmost point of the line, represents no throat pain, and 100mm, the rightmost point of the line, represents the most severe throat pain.

SECONDARY OUTCOMES:
Clinical Efficacy Against Common Cold Symptoms | 48 hours
  Secondary endpoints will include changes to the Modified Jackson Score, measured from Absent=0, Mild=1, Moderate=2 to Severe=3, with a higher score representing worsening of various cold symptoms and a lower score signifying improvement of various cold symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlie Latefi, PhD, Study Director — Applied Biological Laboratories
Locations (6):
- United States (6):
  - Telemedicine and Home Visit, Irvine, California
  - Telemedicine and Home Visit, Washington D.C., District of Columbia
  - Telemedicine and Home Visit, Atlanta, Georgia
  - Telemedicine and Home Visit, Baltimore, Maryland
  - Telemedicine and Home Visit, New York, New York
  - Telemedicine and Home Visit, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Will be determined as needed, if shared no identifiable personal information will be provided.
Supporting Information: Study Protocol, SAP
Time Frame: Will be determined as needed
Access Criteria: Requesting researchers will only receive the participant's code number, age, sex, ethnicity, but no other identifying information.

REFERENCES:
- [Background] Shulman ST, Bisno AL, Clegg HW, Gerber MA, Kaplan EL, Lee G, Martin JM, Van Beneden C. Clinical practice guideline for the diagnosis and management of group A streptococcal pharyngitis: 2012 update by the Infectious Diseases Society of America. Clin Infect Dis. 2012 Nov 15;55(10):1279-82. doi: 10.1093/cid/cis847. PMID 23091044
- [Background] Kim SY, Chang YJ, Cho HM, Hwang YW, Moon YS. Non-steroidal anti-inflammatory drugs for the common cold. Cochrane Database Syst Rev. 2015 Sep 21;2015(9):CD006362. doi: 10.1002/14651858.CD006362.pub4. PMID 26387658
- [Background] Winther B, Gwaltney JM Jr, Mygind N, Turner RB, Hendley JO. Sites of rhinovirus recovery after point inoculation of the upper airway. JAMA. 1986 Oct 3;256(13):1763-7. PMID 3018306
- [Background] Rees GL, Eccles R. Sore throat following nasal and oropharyngeal bradykinin challenge. Acta Otolaryngol. 1994 May;114(3):311-4. doi: 10.3109/00016489409126062. PMID 8073865
- [Background] Proud D, Reynolds CJ, Lacapra S, Kagey-Sobotka A, Lichtenstein LM, Naclerio RM. Nasal provocation with bradykinin induces symptoms of rhinitis and a sore throat. Am Rev Respir Dis. 1988 Mar;137(3):613-6. doi: 10.1164/ajrccm/137.3.613. PMID 3345041
- [Background] Doyle WJ, Boehm S, Skoner DP. Physiologic responses to intranasal dose-response challenges with histamine, methacholine, bradykinin, and prostaglandin in adult volunteers with and without nasal allergy. J Allergy Clin Immunol. 1990 Dec;86(6 Pt 1):924-35. doi: 10.1016/s0091-6749(05)80156-3. PMID 2262647
- [Background] Gupta U, Verma M. Placebo in clinical trials. Perspect Clin Res. 2013 Jan;4(1):49-52. doi: 10.4103/2229-3485.106383. No abstract available. PMID 23533982
- [Background] Schachtel B, Aspley S, Shephard A, Shea T, Smith G, Schachtel E. Utility of the sore throat pain model in a multiple-dose assessment of the acute analgesic flurbiprofen: a randomized controlled study. Trials. 2014 Jul 3;15:263. doi: 10.1186/1745-6215-15-263. PMID 24988909
- [Background] Glatthaar-Saalmuller B, Mair KH, Saalmuller A. Antiviral activity of aspirin against RNA viruses of the respiratory tract-an in vitro study. Influenza Other Respir Viruses. 2017 Jan;11(1):85-92. doi: 10.1111/irv.12421. Epub 2016 Sep 22. PMID 27542891
- [Background] Eccles R, Loose I, Jawad M, Nyman L. Effects of acetylsalicylic acid on sore throat pain and other pain symptoms associated with acute upper respiratory tract infection. Pain Med. 2003 Jun;4(2):118-24. doi: 10.1046/j.1526-4637.2003.03019.x. PMID 12873261
- [Background] Leyva-Grado V, Pugach P, Sadeghi-Latefi N. A novel anti-inflammatory treatment for bradykinin-induced sore throat or pharyngitis. Immun Inflamm Dis. 2021 Dec;9(4):1321-1335. doi: 10.1002/iid3.479. Epub 2021 Jun 21. PMID 34153179
- [Derived] Pugach P, Sadeghi-Latefi N. Supporting respiratory epithelia and lowering inflammation to effectively treat common cold symptoms: A randomized controlled trial. PLoS One. 2024 Nov 27;19(11):e0301959. doi: 10.1371/journal.pone.0301959. eCollection 2024. PMID 39602479

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT06106880/Prot_SAP_001.pdf